CLINICAL TRIAL: NCT04296799
Title: Phase 1, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of SMP-100 in Normal Healthy Volunteers
Brief Title: A Phase 1 Study of SMP-100 in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu SciMount Pharmatech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ChengduSciMount
Record Dates: First submitted 2020-02-26; First posted 2020-03-05 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (Experimental): The study will consist of 6 cohorts (1 cohort per dose level) of 8 subjects (6 subjects receiving the study drug and 2 receiving matching placebo), for a total of 48 subjects.
  Interventions: Drug: SMP-100; Drug: Placebo
- Multiple Ascending Dose (Experimental): The study will consist of 3 cohorts (1 cohort per dose level) of 8 subjects. Six subjects will receive study drug and 2 subjects will receive matching placebo, daily for 14 consecutive days, for a total of 24 subjects (18 study drug; 6 placebo).
  Interventions: Drug: SMP-100; Drug: Placebo

INTERVENTIONS:
Drug: SMP-100 — SAD/MAD
  Other Names: SMP-100 oral solution; ALB-137391(a); CSTI-300
Drug: Placebo — Placebo
  Other Names: Placebo oral solution

SUMMARY:
This will be the first clinical study of oral administration SMP-100 in healthy subjects. The proposed randomized Phase 1 trial is a double-blind, placebo-controlled, single and multiple ascending dose study in approximately 72 healthy male and female subjects.

DETAILED DESCRIPTION:
SMP-100 is a novel serotonin receptor 3 (5-HT3) partial agonist which has been designed to be a safe and effective therapy for irritable bowel syndrome (IBS) patients .

This will be a single center, Phase 1, double-blind, placebo-controlled, randomized, sequential single ascending dose (SAD)/ multiple ascending dose (MAD) study to assess the safety, tolerability, and PK of SMP-100 in healthy adult male and female subjects. The study will be divided into two parts:

Part A: SAD cohorts Part A will consist of 6 cohorts (1 cohort per dose level) of 8 subjects (6 subjects receiving the study drug and 2 receiving matching placebo), for a total of 48 subjects. Each subject will participate in only one cohort. Efforts will be made to randomize at least 3 subjects of each gender in each cohort.

Part B: MAD cohorts Part B will consist of 3 cohorts (1 cohort per dose level) of 8 subjects. Six subjects will receive study drug and 2 subjects will receive matching placebo, daily for 14 consecutive days, for a total of 24 subjects (18 study drug; 6 placebo). Each study subject will participate in only one cohort. Efforts will be made to randomize at least 3 subjects of each gender in each cohort.

For both Part A and Part B, subjects who withdraw or are withdrawn from the study after dosing, for reasons other than safety and tolerability, may be replaced after consultation between the Safety Review Committee (SRC) members. The total number of subjects dosed (including potential replacement subjects) will remain within a maximum of 10 subjects per cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening) aged between ≥18 and ≤59 years old.
2. BMI >18.5 and <30.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
3. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
   3. the absence of clinically significant history of constipation, diarrhea, or irregular bowel transit in the last 4 weeks.
   4. the absence of clinically significant history of irritable bowel syndrome (IBS) of any type.
   5. the absence of current or history of ischemic colitis.
4. Females of childbearing potential who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomized since at least 6 months) must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after (the last) study drug administration:

   1. simultaneous use of intra-uterine contraceptive device placed at least 4 weeks prior to (the first) study drug administration, and condom for the male partner;
   2. simultaneous use of hormonal contraceptive starting at least 4 weeks prior to (the first) study drug administration and must agree to use the same hormonal contraceptive throughout the study, and condom for the male partner;
   3. simultaneous use of diaphragm or cervical cap and male condom for the male partner, started at least 21 days prior to (the first) study drug administration.

   A woman is considered of childbearing potential unless she is surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy) at least 6 weeks before screening or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause).
5. Male subjects who are not vasectomized for at least 6 months, and who are sexually active with a female partner of childbearing potential (childbearing potential females are defined as women that are neither post-menopausal nor surgically sterile) must be willing to use one of the following acceptable contraceptive methods from the first study drug administration until at least 90 days after the last study drug administration:

   1. simultaneous use of a male condom and, for the female partner, hormonal contraceptives used since at least 4 weeks or intra-uterine contraceptive device placed since at least 4 weeks;
   2. simultaneous use of a male condom and, for the female partner, a diaphragm.
6. Male subjects (including men who have had a vasectomy) with a pregnant or same-sex partner must agree to use a condom from the first study drug administration until at least 90 days after the last study drug administration.
7. Male subjects must be willing not to donate sperm until 90 days following the last study drug administration.
8. Willing to take off dentures or mouth piercing at the time of dosing.
9. Capable of consent.

Exclusion Criteria:

1. Any clinically significant abnormality at physical examination.
2. Any clinically significant abnormal laboratory test results or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
3. Positive urine drug screen, alcohol breath test, or urine cotinine test at screening. A repeat test can be conducted at screening or Day -1 at the discretion of the Principal Investigator or delegate.
4. History of allergic reactions to SMP-100 or other related drugs, or to any excipient in the formulation.
5. History of hypersensitivity to 5-HT3 receptor antagonists or agonists.
6. Positive serum pregnancy test at screening.
7. Clinically significant ECG abnormalities (QTcF >450 ms for males and QTcF >460 ms for females).
8. Clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 159 mmHg, diastolic blood pressure lower than 50 or over 100 mmHg, or heart rate less than 50 or over 100 bpm) at screening. Repeat test can be conducted at screening or Day -1 at the discretion of the Principal Investigator or delegate.
9. Clinically significant orthostatic vital sign abnormalities such as decrease in systolic blood pressure of 20 mmHg or higher, decrease in diastolic blood pressure of 10 mmHg or higher, or increase in heart rate of 30 bpm or higher within 3 minutes after passing from a supine to a standing position. Repeat test can be conducted at screening or Day -1 at the discretion of the principal investigator or delegate.
10. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 150 mL of wine, 375 mL of mid strength beer, or 30 mL of 40% alcohol]).
11. History of significant drug abuse within 1 year prior to screening or use of drugs such as marijuana within 3 months prior to the screening visit or drugs such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives within 1 year prior to screening.
12. Participation in a clinical research study involving the administration of an investigational drug or device within 30 days prior to the first dosing.
13. Administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing.
14. Use of medications for the timeframes specified below, with the exception of medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

    1. prescription medications within 14 days prior to the first dosing;
    2. over-the-counter products and natural health products (including herbal remedies homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 14 days prior to the first dosing, with the exception of the occasional use of paracetamol (up to 2 g daily);
    3. any prescription or over-the-counter medication or natural health products used for the treatment of irregular bowel transit (e.g. diarrhea, constipation) within 4 weeks prior to the first dosing;
    4. depot injection or implant of any drug within 3 months prior to the first dosing;
    5. use of any drugs known to induce or inhibit hepatic metabolism (including St. John's Wort [hypericin]) within 14 days prior to the first dosing.
15. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
16. Presence of:

    1. orthodontic braces or orthodontic retention wires, or
    2. any physical findings in the mouth or tongue that would be likely to interfere with successful completion of the dosing procedure.
17. Breast-feeding subject.
18. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Safety Endpoints of SAD | 10±2 days post dose
  Number of subjects with adverse events (AEs) (i.e., seriousness, severity, relationship to the study medication, outcome, duration, and management), vital signs, 12-lead electrocardiogram (ECGs), clinical laboratory parameters, weight, and physical examination.
Safety Endpoints of MAD | 13±2 days post last dose
  Number of subjects with adverse events (AEs) (i.e., seriousness, severity, relationship to the study medication, outcome, duration, and management), vital signs, 12-lead electrocardiogram (ECGs), clinical laboratory parameters, weight, and physical examination.

SECONDARY OUTCOMES:
PK Endpoints AUC0-t of SAD | before dosing and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose.
  area under the concentration-time curve from time zero to the last non-zero concentration (AUC0-t)
PK Endpoints AUC0-24 of SAD | before dosing and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose.
  area under the concentration-time curve from time zero to time 24 hours (AUC0-24)
PK Endpoints AUC0 inf of SAD | before dosing and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose.
  area under the concentration-time curve from time zero to infinity (extrapolated) (AUC0 inf)
PK Endpoints Cmax of SAD | before dosing and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose.
  maximum plasma concentration (Cmax)
PK Endpoints Tmax of SAD | before dosing and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose.
  time of maximum concentration ( Tmax)
PK Endpoints T½ el of SAD | before dosing and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose.
  elimination half-life ( T½ el)
PK Endpoints Cl/F of SAD | before dosing and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose.
  Total body clearance, calculated as Dose / AUC0-inf (Cl/F)
PK Endpoints Vz/F of SAD | before dosing and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours post-dose.
  apparent volume of distribution, calculated as Dose / (Kel * AUC0-inf) (Vz/F)
PK Endpoints AUC0-24 of MAD | Day 1
  area under the concentration-time curve from time zero to time 24 hours (AUC0-24)
PK Endpoints Cmax of MAD | Day 1
  maximum plasma concentration (Cmax)
PK Endpoints Tmax of MAD | Day 1
  time of maximum concentration ( Tmax)
PK Endpoints T½ el of MAD | Day 1
  elimination half-life ( T½ el)
PK Endpoints AUC0-τ of MAD | Day 14
  area under the concentration-time curve at steady-state from time zero to time 24 hours ( AUC0-τ)
PK Endpoints AUC0-48 of MAD | Day 14
  area under the concentration-time curve from time zero to time 48 hours ( AUC0-48)
PK Endpoints AUC0-72 of MAD | Day 14
  area under the concentration-time curve from time zero to time 72 hours ( AUC0-72)
PK Endpoints Cmax ss of MAD | Day 14
  maximum observed concentration at steady-state （Cmax ss）
PK Endpoints Tmax ss of MAD | Day 14
  time of maximum concentration at steady-state（Tmax ss）
PK Endpoints Cmin ss of MAD | Day 14
  minimum observed concentration at steady-state（Cmin ss）
PK Endpoints AUC0- t of MAD | Day 14
  area under the concentration-time curve from time zero to the last non-zero concentration（AUC0- t）
PK Endpoints T½ el of MAD | Day 14
  elimination half-life（T½ el）
PK Endpoints Clss/F of MAD | Day 14
  total body clearance at steady-state, calculated as Dose / AUC0-inf（Clss/F）
PK Endpoints Vz ss/F of MAD | Day 14
  apparent volume of distribution at steady-state, calculated as Dose / (Kel * AUC0-inf)（Vz ss/F）
Plasma concentration observed of MAD | before treatment administrations (Ctrough) during repeated dosing (Days 2-13)
  Plasma concentration observed will be presented

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, Principal Investigator — CMAX Clinical Research Pty Ltd
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, Australia